CLINICAL TRIAL: NCT00305903
Title: A Prospective, 26-Week, Open-Label, Multi-Center, Single-Arm Pilot Study to Evaluate the Safety and Tolerability of Rivastigmine Capsule With Add on Memantine HCl in Patients With Probable Alzheimer's Disease (MMSE 10-20)
Brief Title: Safety and Tolerability of Rivastigmine With Add-on Memantine in Patients With Probable Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CENA713BUS32
Record Dates: First submitted 2006-03-20; First posted 2006-03-22 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Alzheimer's Disease
Keywords: Dementia,; Alzheimer's,; Rivastigmine,; Memantine
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Rivastigmine; Memantine

INTERVENTIONS:
Drug: Rivastigmine, memantine

SUMMARY:
This is a prospective, 26-week, open-label, single-arm multi-center pilot study. Eligible patients will receive open-label treatment with rivastigmine capsules plus memantine tablets as add on therapy. This study is designed to evaluate the safety and tolerability of add on therapy with memantine to rivastigmine capsules in patients with probable AD (MMSE 10-20)

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of probable Alzheimer's disease;
* Have an MMSE score between 10 and 20;
* Must be able to swallow capsule/tablet;
* Must have a caregiver who is able to attend all study visits;

Exclusion Criteria:

* Have an advanced, severe, progressive, or unstable disease of any type that may interfere with efficacy and safety assessments or put the patient at special risk;
* Have a current diagnosis of active, uncontrolled seizure disorder;
* Have a history within the past year or current diagnosis of cerebrovascular disease
* Have a current diagnosis of severe or unstable cardiovascular disease;
* Had a myocardial infarction (MI) within the last six months;
* Have specific respiratory, digestive, renal, or endocrine disorders;
* Have had previous treatment with rivastigmine or memantine;

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-03; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of treatment with memantine and rivastigmine, measured by the incidence of GI adverse events (nausea and vomiting)

SECONDARY OUTCOMES:
Whether patients on rivastigmine and memantine are able to reach and maintain higher doses of rivastigmine compared to historical data of rivastigmine monotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — 862-778-8300
Locations (1):
- Paterson, New Jersey, United States

REFERENCES:
- [Derived] Sadowsky CH, Dengiz A, Meng X, Olin JT; US38 Study Group. Switching from oral donepezil to rivastigmine transdermal patch in Alzheimer's disease: 20-week extension phase results. Prim Care Companion J Clin Psychiatry. 2010;12(5):PCC.09m00852. doi: 10.4088/PCC.09m00852oli. PMID 21274364